CLINICAL TRIAL: NCT02839551
Title: Optimal Step Doses for Drug Provocation Tests to Prove Beta-lactam Hypersensitivity
Brief Title: Optimal Doses for Drug Provocation Tests to Beta-lactams
Acronym: NewBL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL15_0269
Record Dates: First submitted 2016-07-18; First posted 2016-07-21 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2021-12

CONDITIONS: Drug Hypersensitivity
Keywords: Betalactams; Drug hypersensitivity; Drug provocation test; Reactive dose
MeSH Terms: conditions — Drug Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Simplified drug provocation test (Experimental): Assessment of the Hypersensitivity to betalactams by simplified drug provocation test
  Interventions: Procedure: simplified drug provocation test

INTERVENTIONS:
Procedure: simplified drug provocation test — Assessment of the Hypersensitivity to betalactams by simplified drug provocation test

SUMMARY:
Drug provocation tests (DPT) are widely in case of suspicion of drug hypersensitivity (and in the absence of contraindications), but there are no standardized protocols and most groups use hypothesis (clinically-driven) protocols.

investigators used 20 year experience in drug hypersensitivity to analyse retrospectively 171 patients (accounting for 182 positive DPT to beta-lactams). Using survival analysis, they identified optimal doses to include in a data-driven protocol. This data-driven protocol will be applied to new prospective patients, to test its safety and benefits (gain in time, hospital and patient benefits).

ELIGIBILITY:
Inclusion Criteria:

* patients with positive Drug Provocation Test (DPT) to beta-lactams

Exclusion Criteria:

* contra-indications to DPT
* refusal of participation
* vulnerable patients according to French regulation

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1252 (Actual)
Dates: Start 2016-05-04 (Actual); Primary Completion 2021-11-16 (Actual); Study Completion 2021-11-16 (Actual)

PRIMARY OUTCOMES:
Assessment of the new simplified drug provocation test | up to 1 hour
  Assessment of the non inferiority of the new drug provocation test compared to the present drug provocation test

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital of Montpellier, Montpellier, France, France

IPD SHARING:
Plan to Share IPD: Undecided